CLINICAL TRIAL: NCT05249491
Title: Evaluation of the Etiological Factors of Black Tooth Stain in Children
Brief Title: Etiology of Black Tooth Stain in Children
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Dilsah Cogulu, Prof. Dr., Ege University
Other Study IDs: Ege U. Eth. Com.-17-4/18
Record Dates: First submitted 2021-12-20; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2018-12

CONDITIONS: Tooth Discoloration
MeSH Terms: conditions — Tooth Discoloration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Dental plaque samples were collected from cases with black tooth stain and without black stain for microbiological procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Children with black tooth stain
  Interventions: Diagnostic Test: Microbiological evaluation of dental plaques with children with or without black tooth stain
- Group 2: Children without black tooth stain
  Interventions: Diagnostic Test: Microbiological evaluation of dental plaques with children with or without black tooth stain

INTERVENTIONS:
Diagnostic Test: Microbiological evaluation of dental plaques with children with or without black tooth stain — Evaluation of the etiological factors of black tooth stain according to the questionnaire
  Other Names: Etiological factors of black tooth stain

SUMMARY:
The aim of the present study was to investigate the relationship between the presence of black tooth stain (BS) and dental caries incidence, dental plaque scores and to examine the colonization of Streptococcus mutans, Lactobacillus spp., Actinomyces spp. and Capnocytophaga spp. in dental plaque samples with or without BS. The socioeconomic status of the family, the oral hygiene and dietary habits of the children, medical and dental history of the children were also compared between two groups.

DETAILED DESCRIPTION:
A total of 1000 children aged 3-12 years who applied to the Department of Pedodontics, Faculty of Dentistry, Ege University for routine dental examination were enrolled the study. From these group, children with BS (n=44) were selected as the study group. With the same number of the study group, with the same age and same sex, children without BS (n=44) were categorized as the control group. The parents were interviewed based on a structured questionnaire including questions on the socioeconomic status of the family, the oral hygiene and dietary habits of the children, medical and dental history of the children. The presence and grading of BS, dental caries incidence and dental plaque index scores were recorded by the same pediatric dentist (G.İ.). Dental examinations of the children were conducted under natural light with the aid of a dental mirror and explorer. Dental caries scores were recorded according to WHO (World Health Organization) criteria using DMFT/DMFS (decay, missing, filled, tooth/surface in permanent teeth) and dmft/dmfs indices (decay, missing, filled, tooth/surface in primary teeth). All children were classified according to the DMFT/dmft scores; Group-1: caries active (dmft+DMFT≥1), Group-2: caries-free (dmft+DMFT=0). Dental plaque scores were recorded according to Silness & Löe index. The BS scores were classified according to Gasparetto et al. The plaque samples were dispersed in a vortex mixer to obtain a homogeneous suspension and cultivated on selective VCAT medium (Oxoid) for Capnocytophaga spp., mitis salivarius agar (Difco) with 15% sucrose (Difco) and 0.2 units/mL of bacitracin (Sigma, Sigma-Aldrich Co., St Louis, MO, USA) for S. mutans , MRS Agar was used for the isolation of lactobacilli spp. (ref) and Actinomyces Selective Agar was used for the isolation of Actinomyces spp.

All data were analyzed by SPPS 25.0 (SPSS Statistics for Windows, Armonk, NY: IBM Corp.). In the analysis of data, t test and Mann Whitney-U test were used for the comparison of the two groups. Categorical data were analyzed by Fisher's Exact Test and chi square test. For the significance level of the tests, p<0.05 and p<0.01 were accepted.

ELIGIBILITY:
Inclusion Criteria:

* Cooperative children with or without black tooth stain.
* Children aged between 3-12 years old.

Exclusion Criteria:

* Uncooperative children.
* Children who had taken antibiotic therapy within 3 months prior to the dental plaque sampling and children with any systemic disease were not included to the study.
* Children having oral disease (periodontitis, oral mucosal disease etc.)
* Children having autoimmune disease.
* Parents refuse to sign the consent.

Ages: 3 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: 44 children with black tooth stain and 44 children without black tooth stain with the age 3-12 years old.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-06-10 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Salivary bacterial level | 6 months
  Sample collection from dental plaque

SECONDARY OUTCOMES:
Dental caries experience | 6 months
  The dental caries incidence of all patients were recorded according to the dfs, DMFS indices

OTHER OUTCOMES:
Etiological factors of black tooth stain | 6 months
  The etiological factors of black tooth stain was determined according to the structured questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Dilşah Çoğulu, Prof. Dr., Study Director — Ege University, Izmir, Turkey
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No